CLINICAL TRIAL: NCT02948998
Title: Evaluating the Effect of Spironolactone on Hypertrophic Cardiomyopathy-- a Multicenter Randomized Control Trial
Brief Title: Evaluating the Effect of Spironolactone on Hypertrophic Cardiomyopathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Ruijin Hospital (Other); RenJi Hospital (Other); Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XH-16-032
Record Dates: First submitted 2016-10-27; First posted 2016-10-31 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2017-10

CONDITIONS: Hypertrophic Cardiomyopathy; Fibrosis
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Fibrosis | interventions — Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): The participants in control group do not take spironolactone.
- spironolactone (Experimental): The participants in spironolactone group take 10-20mg spironolactone orally and daily.
  Interventions: Drug: Spironolactone

INTERVENTIONS:
Drug: Spironolactone — The participants in this arm will be prescribed to take 20mg spironolactone orally and daily. Serum potassium concentration and creatinine and blood pressure will be monitored regularly to make the participants safe.
  Other Names: LuoNeiZhi
  Arms: spironolactone

SUMMARY:
Hypertrophic Cardiomyopathy (HCM) is the most common hereditary heart disease with high mortality. Heart failure is the most common complication (about 50% incidence) in these patients. However, it is lack of efficiency medicine to treat heart failure for HCM patients.

Recent studies found fibrosis was common in HCM patients and it was progressive with aging. Late gadolinium enhancement cardiac magnetic resonance (LGE-CMR) is a gold standard to measure the left ventricular(LV) fibrosis extent and been proven to be useful in HCM patients.

Aldosterone plays an important role in the development of fibrosis. Meanwhile, a few studies suggested that aldosterone might participate the development of fibrosis in HCM patients. Spironolactone, a mineralocorticoid receptor antagonist, has been proven its effect on inceasing the survival of the heart-failure patients with the eject fraction lower than 35%.

Thus, the investigators hypothesize that fibrosis is one important reason of heart failure for HCM patients. The purpose of this study is to investigate whether small dosage and early prescription of spironolactone to HCM patients can relieve and/or reverse the fibrosis progress and improve patients' symptoms.

This study is a multicenter, randomized, controlled and open-label study being conducted in 4 centers in Shanghai, China. The primary objective of the study is to evaluate the efficacy of spironolactone on relieving the LV fibrosis in HCM patients. This study plans to recruit 260 participants with definite HCM diagnosis. Then these participants will be randomized to two groups-- "control group "(not taking spironolactone) and "spironolactone group" (taking 20mg spironolactone orally and daily). LGE-CMR, echocardiography, 24-hour Holter, electrocardiography (ECG), and blood test (including hemoglobin, creatitine, potassium, liver enzymes, proBNP, TnT, angiotensin and aldosterone) will be performed before random allocation and after 2 years. LGE-CMR will be used to measure the extent of fibrosis in LV. The extent of LGE+% (the area showing LGE divided by the total area) before and after 2-year experiment and the increase of LGE+% after 2-year experiment will be compared between control and spironolactone groups. Meanwhile, symptoms, New York Heart Association classification of cardiac function, arrhythmia, proBNP and TnT etc. will be compared between two groups.

DETAILED DESCRIPTION:
Hypertrophic Cardiomyopathy (HCM) is the most common hereditary heart disease. Approximate 1--2% population of HCM patients die every year because of cardiocerebrovascular complications in which heart failure, stroke and sudden cardiac deaths rank the top three. Among them, heart failure has the highest incidence (about 50%) but the least ways to treat. Even though the Heart Association of United States and Europe updated the guidelines for the diagnosis and management of HCM, it is still lack of qualified clinical trials about medicine for HCM in the real world.

Late gadolinium enhancement cardiac magnetic resonance (LGE-CMR) is a gold standard to measure the left ventricular(LV) fibrosis extent. Recent studies found that: (1)a proportion of HCM patients have LV fibrosis during the early stage of disease; (2)the LV fibrosis in the HCM patients is progressive; (3)about 91.5% population of HCM patients had late gadolinium enhancement; and(4) late gadolinium enchancement in the HCM patients is related to the risk of sudden death.

Fibrosis is an important pathology of heart failure for the patients with coronary artery disease and dilated cardiomyopathy. The activation of renin-angiotensin-aldosterone system plays a key role during the progression of heart failure. Small dosage of spironolactone has been proven its effect on inceasing the survival of the heart-failure patients with the eject fraction lower than 35%. Meanwhile, a few studies found aldosterone levels of LV myocytes increased both in HCM patients and HCM transgenic mice. Furthermore, spironolactone, a mineralocorticoid receptor antagonist, could reserve interstitial fibrosis, attenuate myocyte disarray by 50%, and improve diastolic function in HCM transgenic mice.

Thus, the investigators hypothesize that fibrosis is one important reason of heart failure for HCM patients and small dosage and early prescription of spironolactone to HCM patients can relieve and/or reverse the fibrosis progress and improve patients' symptoms.

This study is a multicenter, randomized, controlled and open-label study being conducted in 4 centers in Shanghai, China. The primary objective of the study is to evaluate the efficacy of spironolactone on relieving the LV fibrosis in HCM patients.

This study plans to recruit 260 participants with definite HCM diagnosis. Then these participants will be randomized to two groups-- "control group "(not taking spironolactone) and "spironolactone group" (taking 20mg spironolactone orally and daily). LGE-CMR, echocardiography, 24-hour Holter, electrocardiography (ECG), and blood test (including hemoglobin, creatitine, potassium, liver enzymes, proBNP, TnT, angiotensin and aldosterone) will be performed before random allocation and after 2 years.

LGE-CMR will be used to measure the extent of fibrosis in LV. Myocardial areas showing signal intensity >5 SD than mean signal intensity of normal myocardium were defined as segments with LGE. LGE extent in each segment was expressed as the surface area showing LGE divided by the total area of the given myocardial segment, and then summation of the planimetered LGE areas in all short-axis slices yielded total LGE extent, which was subsequently expressed as a proportion of total LV myocardium (LGE+%).

The extent of LGE+% before and after 2-year experiment and the increase of LGE+% after 2-year experiment will be compared between control and spironolactone groups. Meanwhile, symptoms, New York Heart Association classification of cardiac function, arrhythmia, proBNP and TnT etc. will be compared between two groups.

ELIGIBILITY:
Inclusion Criteria:

* male or female, aged from 18 to 75 years
* a wall thickness ≥15mm in one or more LV myocardial segments -- as measured by any imaging technique (echocardiography, cardiac magnetic resonance imaging (CMR) or computed tomography (CT) --that is not explained solely by loading conditions
* LVEF≥50%
* serum potassium <5.0mmol/L
* systolic blood pressure ≥100mmHg
* not taking spironolactone for the last 6 months
* willing to comply with scheduled visits
* informed consent form signed by the subject before participation in the trial

Exclusion Criteria:

* cardiac magnetic resonance imaging (CMR) can not be accepted
* spironolactone is not tolerant or is contradicted
* taking spironolactone during the last 6 months
* severe systemic illness with life expectancy judged < 3 years
* expected to have ventricular septal myectomy or septal alcohol ablation during the trial
* expected to have valve repair or replacement during the trial
* history of myocardial infarction
* angiotension-converting-enzyme inhibitor (ACE-I) or AT-1 receptor blockade is obligatory because of any reason
* systolic blood pressure <90mmHg
* known orthostatic hypotension
* history of hyperkalemia (serum potassium ≥5.5mmol/L) in the past 6 months or serum potassium ≥5.0mmol/L within the past 2 weeks
* severe renal dysfunction, defined as an eGFR <30mL/min or serum creatinine ≥221mmol/L
* hemodialysis
* known chronic hepatic disease, defined as aspartate aminotransferase and alanine aminotransferase levels > 3 times the upper limit of normal as read at the local laboratory
* women of child-bearing or lactation
* cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2018-05-14 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
the extent of late gadolinium enhancement (LGE+%) | 2 years
  LGE-CMR will be used to measure the extent of LV fibrosis in the participants. LGE extent in each segment was expressed as the surface area showing LGE divided by the total area of the given myocardial segment, and then summation of the planimetered LGE areas in all short-axis slices yielded total LGE extent, which was subsequently expressed as a proportion of total LV myocardium (%LGE).

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Gang Li, MD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medcine
Locations (1):
- Xinhua Hospital, Shanghai Jiao Tong University School of Medicne, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ammirati E, Contri R, Coppini R, Cecchi F, Frigerio M, Olivotto I. Pharmacological treatment of hypertrophic cardiomyopathy: current practice and novel perspectives. Eur J Heart Fail. 2016 Sep;18(9):1106-18. doi: 10.1002/ejhf.541. Epub 2016 Apr 24. PMID 27109894
- [Background] Semsarian C, Ingles J, Maron MS, Maron BJ. New perspectives on the prevalence of hypertrophic cardiomyopathy. J Am Coll Cardiol. 2015 Mar 31;65(12):1249-1254. doi: 10.1016/j.jacc.2015.01.019. PMID 25814232
- [Background] Maron BJ, Maron MS. The 20 advances that have defined contemporary hypertrophic cardiomyopathy. Trends Cardiovasc Med. 2015 Jan;25(1):54-64. doi: 10.1016/j.tcm.2014.09.004. PMID 25446045
- [Background] Ho CY, Lakdawala NK, Cirino AL, Lipshultz SE, Sparks E, Abbasi SA, Kwong RY, Antman EM, Semsarian C, Gonzalez A, Lopez B, Diez J, Orav EJ, Colan SD, Seidman CE. Diltiazem treatment for pre-clinical hypertrophic cardiomyopathy sarcomere mutation carriers: a pilot randomized trial to modify disease expression. JACC Heart Fail. 2015 Feb;3(2):180-8. doi: 10.1016/j.jchf.2014.08.003. Epub 2014 Oct 31. PMID 25543971
- [Background] Choi HM, Kim KH, Lee JM, Yoon YE, Lee SP, Park EA, Lee W, Kim YJ, Cho GY, Sohn DW, Kim HK. Myocardial fibrosis progression on cardiac magnetic resonance in hypertrophic cardiomyopathy. Heart. 2015 Jun;101(11):870-6. doi: 10.1136/heartjnl-2014-306555. Epub 2015 Apr 20. PMID 25897040
- [Background] Briasoulis A, Mallikethi-Reddy S, Palla M, Alesh I, Afonso L. Myocardial fibrosis on cardiac magnetic resonance and cardiac outcomes in hypertrophic cardiomyopathy: a meta-analysis. Heart. 2015 Sep;101(17):1406-11. doi: 10.1136/heartjnl-2015-307682. Epub 2015 Jun 9. PMID 26060120
- [Background] Maron BJ, Ommen SR, Semsarian C, Spirito P, Olivotto I, Maron MS. Hypertrophic cardiomyopathy: present and future, with translation into contemporary cardiovascular medicine. J Am Coll Cardiol. 2014 Jul 8;64(1):83-99. doi: 10.1016/j.jacc.2014.05.003. PMID 24998133
- [Background] Huang W, Liang J, Kazmierczak K, Muthu P, Duggal D, Farman GP, Sorensen L, Pozios I, Abraham TP, Moore JR, Borejdo J, Szczesna-Cordary D. Hypertrophic cardiomyopathy associated Lys104Glu mutation in the myosin regulatory light chain causes diastolic disturbance in mice. J Mol Cell Cardiol. 2014 Sep;74:318-29. doi: 10.1016/j.yjmcc.2014.06.011. Epub 2014 Jun 30. PMID 24992035
- [Background] Authors/Task Force members; Elliott PM, Anastasakis A, Borger MA, Borggrefe M, Cecchi F, Charron P, Hagege AA, Lafont A, Limongelli G, Mahrholdt H, McKenna WJ, Mogensen J, Nihoyannopoulos P, Nistri S, Pieper PG, Pieske B, Rapezzi C, Rutten FH, Tillmanns C, Watkins H. 2014 ESC Guidelines on diagnosis and management of hypertrophic cardiomyopathy: the Task Force for the Diagnosis and Management of Hypertrophic Cardiomyopathy of the European Society of Cardiology (ESC). Eur Heart J. 2014 Oct 14;35(39):2733-79. doi: 10.1093/eurheartj/ehu284. Epub 2014 Aug 29. No abstract available. PMID 25173338
- [Background] Hamada M, Ikeda S, Shigematsu Y. Advances in medical treatment of hypertrophic cardiomyopathy. J Cardiol. 2014 Jul;64(1):1-10. doi: 10.1016/j.jjcc.2014.02.022. Epub 2014 Apr 13. PMID 24735741
- [Background] Almaas VM, Haugaa KH, Strom EH, Scott H, Smith HJ, Dahl CP, Geiran OR, Endresen K, Aakhus S, Amlie JP, Edvardsen T. Noninvasive assessment of myocardial fibrosis in patients with obstructive hypertrophic cardiomyopathy. Heart. 2014 Apr;100(8):631-8. doi: 10.1136/heartjnl-2013-304923. Epub 2013 Dec 24. PMID 24368281
- [Background] Sherrid MV, Shetty A, Winson G, Kim B, Musat D, Alviar CL, Homel P, Balaram SK, Swistel DG. Treatment of obstructive hypertrophic cardiomyopathy symptoms and gradient resistant to first-line therapy with beta-blockade or verapamil. Circ Heart Fail. 2013 Jul;6(4):694-702. doi: 10.1161/CIRCHEARTFAILURE.112.000122. Epub 2013 May 23. PMID 23704138
- [Background] Moravsky G, Ofek E, Rakowski H, Butany J, Williams L, Ralph-Edwards A, Wintersperger BJ, Crean A. Myocardial fibrosis in hypertrophic cardiomyopathy: accurate reflection of histopathological findings by CMR. JACC Cardiovasc Imaging. 2013 May;6(5):587-96. doi: 10.1016/j.jcmg.2012.09.018. Epub 2013 Apr 10. PMID 23582356
- [Background] Maron BJ, Maron MS. Hypertrophic cardiomyopathy. Lancet. 2013 Jan 19;381(9862):242-55. doi: 10.1016/S0140-6736(12)60397-3. Epub 2012 Aug 6. PMID 22874472
- [Background] Brown NJ. Contribution of aldosterone to cardiovascular and renal inflammation and fibrosis. Nat Rev Nephrol. 2013 Aug;9(8):459-69. doi: 10.1038/nrneph.2013.110. Epub 2013 Jun 18. PMID 23774812
- [Background] Todiere G, Aquaro GD, Piaggi P, Formisano F, Barison A, Masci PG, Strata E, Bacigalupo L, Marzilli M, Pingitore A, Lombardi M. Progression of myocardial fibrosis assessed with cardiac magnetic resonance in hypertrophic cardiomyopathy. J Am Coll Cardiol. 2012 Sep 4;60(10):922-9. doi: 10.1016/j.jacc.2012.03.076. PMID 22935464
- [Background] Spoladore R, Maron MS, D'Amato R, Camici PG, Olivotto I. Pharmacological treatment options for hypertrophic cardiomyopathy: high time for evidence. Eur Heart J. 2012 Jul;33(14):1724-33. doi: 10.1093/eurheartj/ehs150. Epub 2012 Jun 19. PMID 22719025
- [Background] Pasquale F, Syrris P, Kaski JP, Mogensen J, McKenna WJ, Elliott P. Long-term outcomes in hypertrophic cardiomyopathy caused by mutations in the cardiac troponin T gene. Circ Cardiovasc Genet. 2012 Feb 1;5(1):10-7. doi: 10.1161/CIRCGENETICS.111.959973. Epub 2011 Dec 5. PMID 22144547
- [Background] Maron MS, Rowin EJ, Lin D, Appelbaum E, Chan RH, Gibson CM, Lesser JR, Lindberg J, Haas TS, Udelson JE, Manning WJ, Maron BJ. Prevalence and clinical profile of myocardial crypts in hypertrophic cardiomyopathy. Circ Cardiovasc Imaging. 2012 Jul;5(4):441-7. doi: 10.1161/CIRCIMAGING.112.972760. Epub 2012 May 4. PMID 22563033
- [Background] Ho CY, Lopez B, Coelho-Filho OR, Lakdawala NK, Cirino AL, Jarolim P, Kwong R, Gonzalez A, Colan SD, Seidman JG, Diez J, Seidman CE. Myocardial fibrosis as an early manifestation of hypertrophic cardiomyopathy. N Engl J Med. 2010 Aug 5;363(6):552-63. doi: 10.1056/NEJMoa1002659. PMID 20818890
- [Background] Orenes-Pinero E, Hernandez-Romero D, Jover E, Valdes M, Lip GY, Marin F. Impact of polymorphisms in the renin-angiotensin-aldosterone system on hypertrophic cardiomyopathy. J Renin Angiotensin Aldosterone Syst. 2011 Dec;12(4):521-30. doi: 10.1177/1470320311405247. Epub 2011 Apr 20. PMID 21507890
- [Background] Flett AS, Hasleton J, Cook C, Hausenloy D, Quarta G, Ariti C, Muthurangu V, Moon JC. Evaluation of techniques for the quantification of myocardial scar of differing etiology using cardiac magnetic resonance. JACC Cardiovasc Imaging. 2011 Feb;4(2):150-6. doi: 10.1016/j.jcmg.2010.11.015. PMID 21329899
- [Background] American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines; American Association for Thoracic Surgery; American Society of Echocardiography; American Society of Nuclear Cardiology; Heart Failure Society of America; Heart Rhythm Society; Society for Cardiovascular Angiography and Interventions; Society of Thoracic Surgeons; Gersh BJ, Maron BJ, Bonow RO, Dearani JA, Fifer MA, Link MS, Naidu SS, Nishimura RA, Ommen SR, Rakowski H, Seidman CE, Towbin JA, Udelson JE, Yancy CW. 2011 ACCF/AHA guideline for the diagnosis and treatment of hypertrophic cardiomyopathy: executive summary: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Thorac Cardiovasc Surg. 2011 Dec;142(6):1303-38. doi: 10.1016/j.jtcvs.2011.10.019. No abstract available. PMID 22093712
- [Background] Maron BJ, Haas TS, Kitner C, Lesser JR. Onset of apical hypertrophic cardiomyopathy in adulthood. Am J Cardiol. 2011 Dec 15;108(12):1783-7. doi: 10.1016/j.amjcard.2011.07.048. Epub 2011 Sep 28. PMID 21958740
- [Background] Melacini P, Basso C, Angelini A, Calore C, Bobbo F, Tokajuk B, Bellini N, Smaniotto G, Zucchetto M, Iliceto S, Thiene G, Maron BJ. Clinicopathological profiles of progressive heart failure in hypertrophic cardiomyopathy. Eur Heart J. 2010 Sep;31(17):2111-23. doi: 10.1093/eurheartj/ehq136. Epub 2010 May 31. PMID 20513729
- [Background] McLeod CJ, Ackerman MJ, Nishimura RA, Tajik AJ, Gersh BJ, Ommen SR. Outcome of patients with hypertrophic cardiomyopathy and a normal electrocardiogram. J Am Coll Cardiol. 2009 Jul 14;54(3):229-33. doi: 10.1016/j.jacc.2009.02.071. PMID 19589435
- [Background] Rudolph A, Abdel-Aty H, Bohl S, Boye P, Zagrosek A, Dietz R, Schulz-Menger J. Noninvasive detection of fibrosis applying contrast-enhanced cardiac magnetic resonance in different forms of left ventricular hypertrophy relation to remodeling. J Am Coll Cardiol. 2009 Jan 20;53(3):284-91. doi: 10.1016/j.jacc.2008.08.064. PMID 19147047
- [Background] Maron MS, Maron BJ, Harrigan C, Buros J, Gibson CM, Olivotto I, Biller L, Lesser JR, Udelson JE, Manning WJ, Appelbaum E. Hypertrophic cardiomyopathy phenotype revisited after 50 years with cardiovascular magnetic resonance. J Am Coll Cardiol. 2009 Jul 14;54(3):220-8. doi: 10.1016/j.jacc.2009.05.006. PMID 19589434
- [Background] Haghjoo M, Mohammadzadeh S, Taherpour M, Faghfurian B, Fazelifar AF, Alizadeh A, Rad MA, Sadr-Ameli MA. ST-segment depression as a risk factor in hypertrophic cardiomyopathy. Europace. 2009 May;11(5):643-9. doi: 10.1093/europace/eun393. Epub 2009 Jan 22. PMID 19164362
- [Background] Kim JB, Porreca GJ, Song L, Greenway SC, Gorham JM, Church GM, Seidman CE, Seidman JG. Polony multiplex analysis of gene expression (PMAGE) in mouse hypertrophic cardiomyopathy. Science. 2007 Jun 8;316(5830):1481-4. doi: 10.1126/science.1137325. PMID 17556586
- [Background] de Resende MM, Kriegel AJ, Greene AS. Combined effects of low-dose spironolactone and captopril therapy in a rat model of genetic hypertrophic cardiomyopathy. J Cardiovasc Pharmacol. 2006 Dec;48(6):265-73. doi: 10.1097/01.fjc.0000248236.43760.86. PMID 17204904
- [Background] Sherrid MV, Barac I, McKenna WJ, Elliott PM, Dickie S, Chojnowska L, Casey S, Maron BJ. Multicenter study of the efficacy and safety of disopyramide in obstructive hypertrophic cardiomyopathy. J Am Coll Cardiol. 2005 Apr 19;45(8):1251-8. doi: 10.1016/j.jacc.2005.01.012. PMID 15837258
- [Background] Hughes SE. The pathology of hypertrophic cardiomyopathy. Histopathology. 2004 May;44(5):412-27. doi: 10.1111/j.1365-2559.2004.01835.x. PMID 15139989
- [Background] Faber L, Seggewiss H, Welge D, Fassbender D, Schmidt HK, Gleichmann U, Horstkotte D. Echo-guided percutaneous septal ablation for symptomatic hypertrophic obstructive cardiomyopathy: 7 years of experience. Eur J Echocardiogr. 2004 Oct;5(5):347-55. doi: 10.1016/j.euje.2004.01.001. PMID 15341870
- [Background] Tsybouleva N, Zhang L, Chen S, Patel R, Lutucuta S, Nemoto S, DeFreitas G, Entman M, Carabello BA, Roberts R, Marian AJ. Aldosterone, through novel signaling proteins, is a fundamental molecular bridge between the genetic defect and the cardiac phenotype of hypertrophic cardiomyopathy. Circulation. 2004 Mar 16;109(10):1284-91. doi: 10.1161/01.CIR.0000121426.43044.2B. Epub 2004 Mar 1. PMID 14993121
- [Background] Zou Y, Song L, Wang Z, Ma A, Liu T, Gu H, Lu S, Wu P, Zhang dagger Y, Shen dagger L, Cai Y, Zhen double dagger Y, Liu Y, Hui R. Prevalence of idiopathic hypertrophic cardiomyopathy in China: a population-based echocardiographic analysis of 8080 adults. Am J Med. 2004 Jan 1;116(1):14-8. doi: 10.1016/j.amjmed.2003.05.009. PMID 14706660
- [Background] Choudhury L, Mahrholdt H, Wagner A, Choi KM, Elliott MD, Klocke FJ, Bonow RO, Judd RM, Kim RJ. Myocardial scarring in asymptomatic or mildly symptomatic patients with hypertrophic cardiomyopathy. J Am Coll Cardiol. 2002 Dec 18;40(12):2156-64. doi: 10.1016/s0735-1097(02)02602-5. PMID 12505229
- [Background] Maron BJ, Olivotto I, Bellone P, Conte MR, Cecchi F, Flygenring BP, Casey SA, Gohman TE, Bongioanni S, Spirito P. Clinical profile of stroke in 900 patients with hypertrophic cardiomyopathy. J Am Coll Cardiol. 2002 Jan 16;39(2):301-7. doi: 10.1016/s0735-1097(01)01727-2. PMID 11788223
- [Background] Maron BJ, Niimura H, Casey SA, Soper MK, Wright GB, Seidman JG, Seidman CE. Development of left ventricular hypertrophy in adults in hypertrophic cardiomyopathy caused by cardiac myosin-binding protein C gene mutations. J Am Coll Cardiol. 2001 Aug;38(2):315-21. doi: 10.1016/s0735-1097(01)01386-9. PMID 11499718
- [Background] Spirito P, Bellone P, Harris KM, Bernabo P, Bruzzi P, Maron BJ. Magnitude of left ventricular hypertrophy and risk of sudden death in hypertrophic cardiomyopathy. N Engl J Med. 2000 Jun 15;342(24):1778-85. doi: 10.1056/NEJM200006153422403. PMID 10853000
- [Background] Shirani J, Pick R, Roberts WC, Maron BJ. Morphology and significance of the left ventricular collagen network in young patients with hypertrophic cardiomyopathy and sudden cardiac death. J Am Coll Cardiol. 2000 Jan;35(1):36-44. doi: 10.1016/s0735-1097(99)00492-1. PMID 10636256
- [Background] Basso C, Thiene G, Corrado D, Buja G, Melacini P, Nava A. Hypertrophic cardiomyopathy and sudden death in the young: pathologic evidence of myocardial ischemia. Hum Pathol. 2000 Aug;31(8):988-98. doi: 10.1053/hupa.2000.16659. PMID 10987261
- [Background] Varnava AM, Elliott PM, Sharma S, McKenna WJ, Davies MJ. Hypertrophic cardiomyopathy: the interrelation of disarray, fibrosis, and small vessel disease. Heart. 2000 Nov;84(5):476-82. doi: 10.1136/heart.84.5.476. PMID 11040002
- [Background] Pitt B, Zannad F, Remme WJ, Cody R, Castaigne A, Perez A, Palensky J, Wittes J. The effect of spironolactone on morbidity and mortality in patients with severe heart failure. Randomized Aldactone Evaluation Study Investigators. N Engl J Med. 1999 Sep 2;341(10):709-17. doi: 10.1056/NEJM199909023411001. PMID 10471456
- [Background] Maron BJ, Mathenge R, Casey SA, Poliac LC, Longe TF. Clinical profile of hypertrophic cardiomyopathy identified de novo in rural communities. J Am Coll Cardiol. 1999 May;33(6):1590-5. doi: 10.1016/s0735-1097(99)00039-x. PMID 10334429
- [Background] Rosing DR, Kent KM, Maron BJ, Condit J, Epstein SE. Verapamil therapy: a new approach to pharmacologic treatment of hypertrophic cardiomyopathy. Chest. 1980 Jul;78(1 Suppl):239-47. doi: 10.1378/chest.78.1_supplement.239. PMID 6995039
- [Background] Rosing DR, Kent KM, Borer JS, Seides SF, Maron BJ, Epstein SE. Verapamil therapy: a new approach to the pharmacologic treatment of hypertrophic cardiomyopathy. I. Hemodynamic effects. Circulation. 1979 Dec;60(6):1201-7. doi: 10.1161/01.cir.60.6.1201. PMID 574066
- [Background] Anderson KR, Sutton MG, Lie JT. Histopathological types of cardiac fibrosis in myocardial disease. J Pathol. 1979 Jun;128(2):79-85. doi: 10.1002/path.1711280205. PMID 572867